CLINICAL TRIAL: NCT07241949
Title: Paravertebral Block or External Oblique Intercostal Block? A Comparative Analysis of Pain and Opioid Consumption After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Regional Analgesia Techniques for Laparoscopic Cholecystectomy
Acronym: PVB-EOI-PCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Nurefsan Sadikoglu, Attending Specialist, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pending-EC-2025-NSadikoglu
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Laparoscopic Cholecystectomy; Paravertebral Block; External Oblique Intercostal Plane Block; Patient Controlled Analgesia
Keywords: Cholecystectomy; Pain; Analgesia; Tramadol; Nerve Block
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel study arms: (1) paravertebral block, (2) external oblique intercostal block, or (3) intravenous patient-controlled analgesia (PCA) with tramadol. Each participant will receive only the intervention assigned to their group, and no crossover between groups will occur. Outcomes will be assessed over the first 24 postoperative hours following laparoscopic cholecystectomy.
Who Masked: Outcomes Assessor
Masking Description: The investigator assessing postoperative pain scores will be blinded to the intervention group allocation. Patients and anesthesia providers will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paravertebral Block Group (Active Comparator): Participants in this arm will receive bilateral paravertebral block after induction of general anesthesia. Under ultrasound guidance, 0.25% bupivacaine (20 mL per side; total 40 mL) will be administered to provide postoperative analgesia following laparoscopic cholecystectomy. Patients will also receive standard intravenous paracetamol postoperatively.
  Interventions: Procedure: Paravertebral Block (PVB)
- External Oblique Intercostal Block Group (Active Comparator): Participants in this arm will receive bilateral external oblique intercostal (EOI) block after induction of general anesthesia. Under ultrasound guidance, 0.25% bupivacaine (20 mL per side; total 40 mL) will be injected into the fascial plane between the external oblique and intercostal muscles. Standard intravenous paracetamol will be administered postoperatively.
  Interventions: Procedure: External Oblique Intercostal Block (EOI Block)
- Control Group - IV PCA Tramadol (Active Comparator): Participants in this arm will receive intravenous patient-controlled analgesia (PCA) with tramadol for postoperative pain management. The PCA pump will be set to a maximum dose of 400 mg tramadol in 24 hours. Standard intravenous paracetamol (1 g every 8 hours) will also be administered. No regional anesthesia block will be performed in this group.
  Interventions: Drug: Tramadol IV Patient-Controlled Analgesia (PCA)

INTERVENTIONS:
Procedure: Paravertebral Block (PVB) — Ultrasound-guided bilateral thoracic paravertebral block performed after induction of general anesthesia using 0.25% bupivacaine, 20 mL per side (total 40 mL).
  Arms: Paravertebral Block Group
Procedure: External Oblique Intercostal Block (EOI Block) — Ultrasound-guided bilateral external oblique intercostal block performed after induction of general anesthesia with 0.25% bupivacaine, 20 mL per side (total 40 mL), injected between the external oblique and intercostal muscles.
  Arms: External Oblique Intercostal Block Group
Drug: Tramadol IV Patient-Controlled Analgesia (PCA) — Intravenous patient-controlled analgesia (PCA) programmed to deliver tramadol with a maximum dose of 400 mg in 24 hours. Standard analgesia protocol includes IV paracetamol 1 g every 8 hours.
  Other Names: Control group
  Arms: Control Group - IV PCA Tramadol

SUMMARY:
This single-center, prospective, randomized controlled trial aims to compare the effects of paravertebral block (PVB), external oblique intercostal (EOI) block, and intravenous patient-controlled analgesia (PCA) with tramadol on postoperative pain and opioid consumption in patients undergoing elective laparoscopic cholecystectomy. The primary endpoint is total tramadol consumption within 24 hours postoperatively. Secondary outcomes include pain scores, additional analgesic use, incidence of nausea/vomiting, mobilization time, and length of hospital stay.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled clinical trial aims to compare the analgesic efficacy and opioid-sparing effects of paravertebral block (PVB), external oblique intercostal (EOI) block, and intravenous patient-controlled analgesia (IV PCA) in adult patients undergoing elective laparoscopic cholecystectomy (LC) under general anesthesia.

Although laparoscopic cholecystectomy is a minimally invasive procedure, postoperative pain remains a significant clinical problem, particularly during the first 24 hours after surgery. Effective multimodal analgesia is essential to improve patient comfort, facilitate early mobilization, and reduce opioid-related side effects. Regional anesthesia techniques, such as PVB and EOI block, target both somatic and visceral components of pain and may offer superior postoperative analgesia compared with systemic opioid administration alone.

After obtaining informed consent, eligible patients (aged 18-65 years, ASA I-III) scheduled for elective LC will be randomly assigned to one of three groups using the sealed envelope method:

Group P (Paravertebral Block): After induction of general anesthesia, bilateral paravertebral blocks will be performed at thoracic levels with 0.25% bupivacaine (20 mL per side; total 40 mL).

Group E (External Oblique Intercostal Block): After induction, bilateral EOI blocks will be performed using 0.25% bupivacaine (20 mL per side; total 40 mL) injected into the fascial plane between the external oblique and intercostal muscles under ultrasound guidance.

Group C (Control): Patients will receive standard general anesthesia followed by IV PCA with tramadol (maximum dose 400 mg/24h) and IV paracetamol 1 g every 8 hours.

All patients will receive standard intraoperative monitoring and anesthesia management. Postoperative analgesia will be evaluated using an 11-point Numerical Rating Scale (NRS, 0-10) both at rest and during movement at 20 minutes, 6 hpurs, 12 hours, and 24 hours after surgery. If the NRS score is ≥4 in the postoperative care unit, IV morphine (0.05 mg/kg), If the NRS score is ≥7 Meperidine 0.3 mg/kg will be administered as rescue analgesia.

The primary outcome is total tramadol consumption within the first 24 postoperative hours.

Secondary outcomes include pain scores at predefined time points, requirement for rescue analgesics, incidence of postoperative nausea and vomiting (PONV), time to mobilization, and length of hospital stay.

Patients will be followed for 24 hours postoperatively. The anesthesia team performing the blocks will not participate in data collection. Pain assessments will be conducted by an investigator blinded to group allocation to minimize bias.

This study will provide comparative data on two ultrasound-guided regional anesthesia techniques and systemic opioid-based analgesia for LC, aiming to identify the method that ensures optimal postoperative pain control with the least opioid requirement and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Scheduled for elective laparoscopic cholecystectomy under general anesthesia
* ASA physical status I-III
* Able to understand the study procedure and provide informed consent

Exclusion Criteria:

Patient refusal or inability to provide informed consent

Allergy or contraindication to local anesthetics, tramadol, or study medications

Coagulopathy or current anticoagulant therapy

Local infection at the planned block injection site

Severe hepatic or renal impairment

Chronic opioid use or opioid dependence

Neurological or psychiatric disorders affecting pain perception or communication

Pregnancy or breastfeeding

Body mass index (BMI) > 35 kg/m²

Conversion to open cholecystectomy during surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
24-hour postoperative tramadol consumption | Within the first 24 hours after surgery.
  Total amount of intravenous tramadol administered via PCA within the first 24 hours after surgery.

SECONDARY OUTCOMES:
Postoperative pain scores at rest | 1, 6, 12, and 24 hours postoperatively
  Pain intensity at rest assessed using a Numeric Rating Scale (0-10).
Incidence of postoperative nausea and vomiting | Within 24 hours postoperatively
  Presence of nausea and/or vomiting requiring antiemetic treatment.
Incidence of block-related complications | Intraoperative and first 24 hours after block
  Presence of complications related to the regional block (e.g., vascular puncture, pneumothorax, local anesthetic systemic toxicity).
Patient satisfaction with analgesia | 24 hours postoperatively
  Patient-reported satisfaction score for pain management (0 = very dissatisfied, 10 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Nurefsan Sadikoglu, MD, Principal Investigator — Cukurova University Hospital
Locations (1):
- Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in publications (de-identified dataset including primary and secondary outcome variables) will be shared. No information that could identify participants will be included. Data dictionaries and statistical codes may also be made available upon reasonable request for academic and research purposes. Access will be granted after publication and following institutional data-sharing agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data will be available beginning 6-12 months after publication of the primary results and for a period of up to 3 years thereafter.
Access Criteria: Researchers seeking access to the data will be required to submit a methodologically sound proposal and sign a data-use agreement to ensure confidentiality and compliance with ethical standards. Requests will be evaluated by the study investigators and relevant institutional authorities.

REFERENCES:
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Erskine RN, White L. "A review of the external oblique intercostal plane block - a novel approach to analgesia for upper abdominal surgery". J Clin Anesth. 2022 Nov;82:110953. doi: 10.1016/j.jclinane.2022.110953. Epub 2022 Aug 19. No abstract available. PMID 35994942
- [Background] Hamilton DL, Manickam BP, Wilson MAJ, Abdel Meguid E. External oblique fascial plane block. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100256. doi: 10.1136/rapm-2018-100256. Online ahead of print. No abstract available. PMID 30635518
- [Background] Hamilton DL, Manickam BP. Is a Thoracic Fascial Plane Block the Answer to Upper Abdominal Wall Analgesia? Reg Anesth Pain Med. 2018 Nov;43(8):891-892. doi: 10.1097/AAP.0000000000000838. No abstract available. PMID 30339615
- [Background] Kus A, Gurkan Y, Arslan ZI, Akgul AG, Aksu C, Toker K, Solak M. [Our ultrasound-guided paravertebral block experiences in thoracic surgery]. Agri. 2015;27(3):139-42. doi: 10.5505/agri.2015.59885. Turkish. PMID 26356102
- [Background] Barazanchi AWH, MacFater WS, Rahiri JL, Tutone S, Hill AG, Joshi GP; PROSPECT collaboration. Evidence-based management of pain after laparoscopic cholecystectomy: a PROSPECT review update. Br J Anaesth. 2018 Oct;121(4):787-803. doi: 10.1016/j.bja.2018.06.023. Epub 2018 Aug 7. PMID 30236241
- [Background] O'Donovan B, Martin B. The Novel Use of an External Oblique Nerve Catheter After Open Cholecystectomy. Cureus. 2021 Feb 26;13(2):e13580. doi: 10.7759/cureus.13580. PMID 33796423
- [Background] Alper I, Ulukaya S, Yuksel G, Uyar M, Balcioglu T. Laparoscopic cholecystectomy pain: effects of the combination of incisional and intraperitoneal levobupivacaine before or after surgery. Agri. 2014;26(3):107-12. doi: 10.5505/agri.2014.42650. PMID 25205408
- [Background] Shrestha BB, Lakhe G, Ghimire P. Postoperative Pain after Laparoscopic Cholecystectomy in a Tertiary Care Center: A Descriptive Cross-sectional Study. JNMA J Nepal Med Assoc. 2024 Jul 31;62(276):502-506. doi: 10.31729/jnma.8719. PMID 39369396
- [Background] De Cassai A, Sella N, Geraldini F, Tulgar S, Ahiskalioglu A, Dost B, Manfrin S, Karapinar YE, Paganini G, Beldagli M, Luoni V, Ordulu BBK, Boscolo A, Navalesi P. Single-shot regional anesthesia for laparoscopic cholecystectomies: a systematic review and network meta-analysis. Korean J Anesthesiol. 2023 Feb;76(1):34-46. doi: 10.4097/kja.22366. Epub 2022 Nov 8. PMID 36345156